CLINICAL TRIAL: NCT04699474
Title: Protocol for Rapid Onset of Mobilization in Patients With Traumatic Spinal Cord Injury (PROMPT-SCI)
Brief Title: Protocol for Rapid Onset of Mobilization in Patients With Traumatic Spinal Cord Injury
Acronym: PROMPT-SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Collaborators: University of Louisville (Other); Université de Montréal (Other); The Craig H. Neilsen Foundation (Other); École de technologie supérieure (Unknown)
Responsible Party: Principal Investigator, Jean-Marc Mac-Thiong, Principal Investigator, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-1901
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Early in-bed leg cycling (Experimental)
  Interventions: Device: Leg ergometer

INTERVENTIONS:
Device: Leg ergometer — Leg cycling in bed using motorized ergometer

SUMMARY:
PROMPT-SCI (Protocol for Rapid Onset of Mobilization in Patients with Traumatic SCI) is a single-site single-arm proof-of-concept trial. Forty-five patients aged 18 years or older who have sustained a severe traumatic SCI (American Spinal Injury Association Impairment Scale grade A, B or C) from C0 to L1 and undergoing spinal surgery within 48 hours of the injury will be included. Participants will receive daily 30-minute sessions of in-bed leg cycling for 14 consecutive days, initiated within 48 hours after spinal surgery. The feasibility outcomes consist of the 1) absence of serious adverse events associated with cycling sessions, 2) completion of at least 1 full session within 48 hours after spinal surgery for at least 90% of participants, and 3) completion of at least 11 sessions for at least 80% of participants. Patient outcomes 6 weeks and 6 months after injury will be measured from neurofunctional assessments, quality of life questionnaires and inpatient length of stay. Feasibility and patient outcomes will be analysed with descriptive statistics. Patient outcomes will also be compared to a matched historical cohort not receiving in-bed cycling.

ELIGIBILITY:
Inclusion Criteria:

* Blunt traumatic spinal cord injury
* Neurological level of injury from C0 to L2
* American Spinal Injury Association impairment scale grade A, B or C
* Spine surgery performed within 48 hours of injury

Exclusion Criteria:

* Condition limiting patient's ability to engage into cycling
* Medical condition that might interfere with patient's safety if cycling
* Moderate or severe brain injury
* Inability to walk independently prior to injury
* Pre-existing neurological disorder
* Complete spinal cord transection
* Unwilling or unable to comply with scheduled follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Ambulation | 6 months
  Independent walking (with or without device)

SECONDARY OUTCOMES:
Neurological recovery | 6 months
  International Standards for Neurological Classification of Spinal Cord Injury
Function | 6 months
  Spinal Cord Independence Measure
Spasticity | 6 months
  Spinal Cord Assessment Tool for Spastic Reflexes
Health related quality of life | 6 months
  Short-form 36 and World Health Organization Quality of Life - BREF

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc Mac-Thiong, MD, PhD, Principal Investigator — Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Locations (1):
- Hopital du Sacre-Coeur de Montreal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
In line with the recommendations from the Committee on strategies for Responsible Sharing of Clinical Trial Data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Mac-Thiong JM, Richard-Denis A, Petit Y, Bernard F, Barthelemy D, Dionne A, Magnuson DSK. Protocol for rapid onset of mobilisation in patients with traumatic spinal cord injury (PROMPT-SCI) study: a single-arm proof-of-concept trial of early in-bed leg cycling following acute traumatic spinal cord injury. BMJ Open. 2021 Nov 1;11(11):e049884. doi: 10.1136/bmjopen-2021-049884. PMID 34725077